CLINICAL TRIAL: NCT02794077
Title: Metronomic Oral Cyclosphosphamide as Third-line Systemic Treatment or Beyond in Patients With Inoperable Locoregionally Advanced Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Cyclophosphamide for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Victor H.F. Lee, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cyclophosphamide
Record Dates: First submitted 2016-05-30; First posted 2016-06-08 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Recurrent Nasopharyngeal Undifferentiated Carcinoma; Stage IV Nasopharyngeal Undifferentiated Carcinoma
Keywords: Nasopharyngeal undifferentiated carcinoma
MeSH Terms: interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cyclophosphamide (Experimental): Patients receive oral cyclophosphamide 50 to 150mg daily continuously in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide — Patient receive oral cyclophosphamide 50 to 150mg daily continuously in the absence of disease progressive or unacceptable toxicity.
  Other Names: Endoxan

SUMMARY:
There is no standard third-line systemic treatment for inoperable locoregionally advanced recurrent or metastatic nasopharyngeal carcinoma (NPC). We investigated the efficacy and safety of metronomic oral cyclophosphamide as third-line treatment or beyond.

DETAILED DESCRIPTION:
NPC is endemic in Southern China including Hong Kong. Despite aggressive definitive chemoradiotherapy for locoregionally advanced disease, still about 30% develop relapse locoregionally or distally. Salvage or second-course radical radiotherapy with or without chemotherapy may achieve durable disease control for locoregionally advanced recurrent disease. However for those who had received 2 courses of radical radiotherapy or those with distant metastases, systemic chemotherapy would be the only drug of choice. Platinum-based doublet chemotherapy including cisplatin + 5-fluorouracil, capecitabine, gemcitabine or taxane is considered the standard first-line treatment. For second-line treatment, whether platinum-based chemotherapy was given previously is a consideration. Re-challenge with cisplatin and 5-fluorouracil can be considered in patients who enjoyed a good initial response to the same regimen with an intervening disease-free period of more than 1 year.However so far there has been no recognized standard third-line systemic treatment. Metronomic oral chemotherapy may provide an ideal choice patients treated in this setting by shifting the targets from tumor cells to tumor vasculature so as to reduce the chance of drug resistance as well as offering a relatively low toxicity profile to them who have been significantly jeopardized by the long-term complications brought prior courses of radiation therapy, surgery and chemotherapy.

In view of the above, we investigated metronomic open-label oral cyclophosphamide as third-line treatment or beyond in patients with inoperable locoregionally advanced recurrent or metastatic NPC who had failed at least 2 lines of prior systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Inoperable locoregionally advanced recurrent NPC of undifferentiated type beyond curative surgical resection or second and subsequent courses of radical radiotherapy or metastatic disease who all had received at least 2 lines palliative systemic chemotherapy
* Adequate hematological function defined as absolute neutrophil count ≥1.5 × 10^9/l; hemoglobin ≥9.0 g/dl and platelet ≥100 × 10^9/l
* Adequate renal function defined as serum creatinine ≤1.5 × upper normal limit
* Adequate hepatic function defined as serum bilirubin ≤1.5 × upper normal limit; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 × upper normal limit for patients without liver metastases or ≤5 × upper normal limit for those with liver metastases
* Measurable disease according to the RECIST criteria (version 1.1), for the evaluation of measurable disease

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 3 or above
* Known brain metastases or leptomeningeal metastases; Note: symptomatic, and/or if they require immunosuppressive doses of corticosteroids (e.g. > 10 mg/day prednisone or equivalents) for at least 2 weeks prior to study drug administration; patients with treated brain metastases who are deemed clinically stable and without radiological progression on positron emission tomography (PET), MRI or computed tomography (CT) scan performed =< 8 weeks of study entry, are not excluded; Note: primary nasopharyngeal cancers that directly invade the skull base and extend into the infratemporal fossa (e) are not regarded as brain metastases and are not excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cyclophosphamide
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following:
* Pregnant women
* Nursing women
* Men or women of childbearing potential who are unwilling to employ adequate contraception Note: breastfeeding should be discontinued if the mother is treated with cyclophosphamide; women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; they must adhere to contraception for a period of 31 weeks after the last dose of cyclophosphamide
* For patients with unknown human immunodeficiency virus (HIV) status at the time of enrollment, HIV serology must be tested during screening; patients who are tested positive for HIV could be included if there is an adequate cluster of differentiation 4 (CD4) count (> 350/ul) on a stable regimen of highly active anti-retroviral therapy (HAART) with no detectable or minimal viral burden, and no active infections
* Those who cannot provide written informed consent

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2008-01; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 12 months
  Interval between the date of commencement of cyclophosphamide to the date of radiologically confirmed progressive disease or death, whichever comes earlier.

SECONDARY OUTCOMES:
Objective response rate | 12 months
  The percentage of patients who demonstrate complete response or partial response after study medication as assessed by RECIST 1.1
Disease control rate | 12 months
  The percentage of patients who demonstrate complete response, partial response or stable disease after study medication as assessed by RECIST 1.1
Number of participants with treatment-related adverse events as assessed by CTCAE version 4.0 | 12 months
  All treatment-related adverse events as assessed by CTCAE version 4.0 will be recorded
Overall survival | 36 months
  Time interval between the date of commencement of cyclophosphamide to the date of death

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lee, MD, Principal Investigator — Department of Clinical Oncology, The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan for to make individual participant data available.